CLINICAL TRIAL: NCT04287712
Title: Detection of Early-stage Lung Cancer Using Machine Learning and Plasma Metabolomics
Brief Title: Detection of Lung Cancer by Plasma Lipids
Acronym: ELAID
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other); Jiangsu Cancer Institute & Hospital (Other); Peking University Health Science Center (Other)
Responsible Party: Principal Investigator, Jun Wang, Prof, Peking University People's Hospital
Other Study IDs: 2018PHB233-01
Record Dates: First submitted 2020-02-13; First posted 2020-02-27 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Early-Stage Lung Cancer
Keywords: Early-Stage Lung Cancer; Plasma Metabolomics; Lipids; Machine Learning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For enrolled participants, 4 ml of peripheral blood were collected in tubes containing EDTA and all participants had fasted at least 8 hr before blood collection. Whole blood was centrifuged at 1600 g for 10 min followed by centrifugation at 16000 g for 10 min. Plasma aliquots were transferred into cryovials and stored at -80 °C.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants received surgery: Patients who underwent surgery at the Department of Thoracic Surgery of Peaking University People's Hospital, Jiangsu Cancer Hospital, and Beijing Haidian Hospital were enrolled with the following criteria: 1) pathologically confirmed lung cancer; 2) no history of other malignancies; 3) no anti-cancer treatment (chemotherapy, radiotherapy, targeted therapy, etc.) before surgery. Plasma samples were collected before surgery and plasma lipids were detected by mass spectrometry. Pathological diagnosis and clinical characteristics of enrolled participants were retrieved.
  Interventions: Diagnostic Test: Plasma lipids

INTERVENTIONS:
Diagnostic Test: Plasma lipids — Plasma lipids were detected by an Ultimate 3000 ultra-high-performance liquid chromatography (UHPLC) system coupled with Q-Exactive MS (Thermo Scientific) . Then a detection model was built based on plasma lipids using machine learning algorithm.

SUMMARY:
There are no reliable blood-based tests currently available for early-stage lung cancer diagnosis. We try to establish a highly accurate method for detecting early-stage lung cancer by combining machine learning with untargeted and targeted metabolomics .

DETAILED DESCRIPTION:
All plasma lipids were first detected by untargeted metabolomics methods and 9 feature lipids of early-stage lung cancer were selected by support vector machine algorithm. Then, a targeted metabolomics method was developed to detect the 9 lipids quantitatively based on multiple reaction monitoring mode. Finally, a detection model was established based on the 9 lipids.

ELIGIBILITY:
Inclusion Criteria:

1. pulmonary nodules or opacity
2. plan to receive surgery

Exclusion Criteria:

1. history of other malignancies
2. received anti-cancer treatment (chemotherapy, radiotherapy, targeted therapy, etc.) before surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who with pulmonary nodules or opacity and underwent surgery at the Department of Thoracic Surgery of Peaking University People's Hospital, Jiangsu Cancer Hospital, and Beijing Haidian Hospital were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Plasma Lipids | All samples were detected together after participants recruitment and sample collection. All samples were detected within 18 months from sample collection.
  A detection model based on 9 lipids were developed, including 3 lysophosphatidylcholines, 5 phosphatidylcholines, and a triglyceride. The 9 lipids were detected by targeted metabolomics by mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China